CLINICAL TRIAL: NCT00368004
Title: Family Studies of Uveal Coloboma
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060230; 06-EI-0230
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-15

CONDITIONS: Coloboma
Keywords: Coloboma; Genetics; Optic Nerve Coloboma; Chorioretinal Coloboma; Iris Coloboma; Uveal Coloboma
MeSH Terms: conditions — Coloboma; Coloboma of optic nerve

SUMMARY:
This study will identify the genes responsible for uveal coloboma, an abnormal development of the eye caused by incomplete closure of a normally-occurring gap in the eye (the optic fissure) after the fifth week of life in a human embryo. There have been studies of families in which more than one person has been affected by this disorder. Coloboma occurs in about 1 of 10,000 live births and may cause significant vision loss. Researchers seek a better understanding of the genes responsible for this disorder.

Adults and children who have more than one member of the family with uveal coloboma may be eligible for this study. Patients will undergo a detailed medical history and eye examination appropriate for their age. The pupils will be dilated, through the use of eye drops. Dilation will continue for 4 to 6 hours, and wearing of sunglasses can reduce temporary glare that many patients may experience in brightly lit areas. In addition, pictures will be taken of the front or back of the eye, a procedure that also involves dilation of the pupils. Patients who have coloboma will undergo a complete physical examination. Blood samples will be collected, with a total of about 2 tablespoons from patients ages 10 and older and about 1 teaspoon for each 5 pounds of body weight for younger patients. Also, patients with coloboma may be asked to undergo X-rays , ultrasound, or other tests that are medically indicated.

To have enough DNA to study, the researchers may create a cell line to grow more DNA. Laboratory samples will be coded so that there is no identifying information about participants in this study. No other testing or research will be done on blood samples collected unless patients give permission. The researchers will not provide information about patients' health to other people without your express permission.

DETAILED DESCRIPTION:
Objective: To describe phenotypes and find genes causing a developmental and potentially blinding eye condition, uveal coloboma.

Study population: Families where more than one family member has uveal coloboma. Both affected and genetically informative, unaffected members of the family will be recruited.

Design: Observational study.

Outcome measures: Clinical examination, genetic mapping and mutation identification.

ELIGIBILITY:
* This study will enroll 120 adult and children members of families where more than one individual is reported to have coloboma. Affected and unaffected family members will be both enrolled.

INCLUSION CRITERIA:

1. The participant must have any recognizeable form of inherited coloboma.
2. The participant must be a genetically informative member of a family where more than one person is affected by typical uveal coloboma.
3. The participant must be able to comply with the protocol and provide a blood sample.

EXCLUSION CRITERIA:

1. The participant has any syndromic form of coloboma likely due to mutations in a known gene.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-07-28; Study Completion 2013-04-15

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maumenee IH, Mitchell TN. Colobomatous malformations of the eye. Trans Am Ophthalmol Soc. 1990;88:123-32; discussion 133-5. No abstract available. PMID 2095017
- [Background] Ravine D, Ragge NK, Stephens D, Oldridge M, Wilkie AO. Dominant coloboma-microphthalmos syndrome associated with sensorineural hearing loss, hematuria, and cleft lip/palate. Am J Med Genet. 1997 Oct 17;72(2):227-36. doi: 10.1002/(sici)1096-8628(19971017)72:23.0.co;2-p. PMID 9382148
- [Background] Zlotogora J, Legum C, Raz J, Merin S, BenEzra D. Autosomal recessive colobomatous microphthalmia. Am J Med Genet. 1994 Feb 1;49(3):261-2. doi: 10.1002/ajmg.1320490302. PMID 8209881